CLINICAL TRIAL: NCT07017413
Title: Predictors For Transosseous Maxillary Sinus Lift Complications: A Prospective Cohort Study
Brief Title: Predictors For Transosseous Maxillary Sinus Lift Complications
Acronym: PMSL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mustafa Faisal Al-Jamal, BDS, MSc OMFS, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1045125
Record Dates: First submitted 2025-05-25; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Sinus Lift Surgery Complications; Maxillary Sinus Elevation
Keywords: Transosseous sinus lift; Versah sinus lift; Schneiderian membrane perforation; Residual bone height RBH; Maxillary sinus; Densah bur; Implant surgery complications; Risk predictors sinus elevation; MSSM; decision tree

STUDY DESIGN:
Intervention Model Description: All enrolled patients will undergo transosseous maxillary sinus lift using the Versah Densah bur technique. Outcomes and predictors of intraoperative and postoperative complications will be assessed within this cohort.
Masking Description: No masking is used as both the clinician and the patient are aware of the intervention being performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transosseous Sinus Lift Group (Experimental): Patients will undergo transcrestal maxillary sinus lift using the Versah® osseodensification technique. This arm aims to evaluate the predictors of surgical complications, including residual bone height (RBH), maxillary sinus ostium (MSO) status, Schneiderian membrane thickness, surgical site (tooth location), and amount of vertical lifting required.
  Interventions: Procedure: Transosseous Maxillary Sinus Lift using Osseodensification

INTERVENTIONS:
Procedure: Transosseous Maxillary Sinus Lift using Osseodensification — A surgical procedure utilizing the Versah® osseodensification technique for transcrestal sinus floor elevation. The approach involves the use of specialized Densah® burs to prepare the osteotomy and elevate the sinus membrane through a transosseous (crestal) access, avoiding the lateral window technique. No grafting materials will be used in this procedure.

SUMMARY:
This prospective cohort study aims to identify clinical and anatomical predictors for complications following transosseous maxillary sinus lift procedures using the Versah (Densah burs) technique. The study focuses on patients undergoing transcrestal sinus floor elevation without a lateral window, with or without simultaneous dental implant placement. Variables such as residual bone height, sinus membrane thickness, bone density, and patient-related factors are being evaluated. The objective is to enhance risk stratification and optimize treatment planning for transosseous sinus augmentation.

DETAILED DESCRIPTION:
This prospective cohort study investigates potential predictors of complications associated with transosseous sinus lift procedures utilizing the Versah Densah burs technique. Unlike the traditional lateral approach, this method enables internal sinus floor elevation through a crestal access, minimizing invasiveness while allowing for controlled vertical augmentation.

The study population includes partially edentulous patients in need of vertical ridge augmentation in the posterior maxilla. The following parameters are evaluated as possible predictors of intraoperative and postoperative complications:

1. Residual Bone Height (RBH): Measured from the alveolar crest to the sinus floor.
2. Maxillary Sinus Ostium (MSO) Patency: Assessed radiographically to determine if ostial obstruction contributes to sinus-related events.
3. Schneiderian Membrane Thickness: Measured preoperatively via CBCT, as thicker or thinner membranes may influence perforation risk.
4. Surgical Site Location: Categorized based on the involved maxillary posterior region (e.g., premolar vs. molar).
5. Amount of Vertical Lifting: The total height gained through osteotome-mediated or Densah bur-mediated elevation is recorded.

Primary outcome measures include intraoperative membrane perforation, postoperative sinusitis, implant failure, and the need for revision surgery. The study aims to establish reliable preoperative indicators to stratify complication risk, facilitate clinical decision-making, and improve patient outcomes in transosseous sinus elevation procedures.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients requiring dental implants in the posterior maxilla with a residual bone height of < 6 mm.

  2- Good general health and absence of systemic conditions affecting bone healing (e.g., uncontrolled diabetes, osteoporosis).

  3- No history of chronic sinusitis or other significant sinus pathologies

Exclusion Criteria:

* 1- Severe periodontal disease. 2- Residual bone height > 6 mm. 3- History of previous sinus lift procedures or other maxillofacial surgeries. 4- Smokers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of maxillary sinus membrane perforation and graft displacement, and identification of associated predictors | Intraoperative phase to 1 month post-surgery
  This primary outcome assesses the intraoperative occurrence of Schneiderian membrane perforation and graft displacement during transosseous maxillary sinus lift. It also involves the identification of anatomical and surgical predictors, including residual bone height (RBH), maxillary sinus ostium patency, sinus membrane thickness, surgical site, and the amount of vertical lift performed.

SECONDARY OUTCOMES:
Postoperative Infection Rate | Within 3 months postoperatively
  Incidence of infection or sinusitis following the transcrestal sinus lift procedure, confirmed clinically or radiographically.

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - College of Dentistry , University of Baghdad, Baghdad, Bab Almodaum
  - Planto clinic, Baghdad, Mansour

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations and to maintain patient confidentiality. Data will only be used for the purposes of this study and will not be made publicly available.

REFERENCES:
- [Result] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT07017413/Prot_SAP_000.pdf